CLINICAL TRIAL: NCT05721430
Title: Urdu Translation and Cross Cultural Validation of PedsQL Inventory Infant Scale Parent Report Ages 1 to 12 Months
Brief Title: Urdu Translation and Cross Cultural Validation of PedsQL Inventory Infant Scale Parent Report 1 to 12 Months
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Muhammad Asif Javed, Assistant Professor, Riphah International University
Other Study IDs: saiqaT
Record Dates: First submitted 2023-01-31; First posted 2023-02-10 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Infant Development
Keywords: Health related quality of life of Infants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current study aimed to translate and validate Urdu version of that module from PedsQL, to measure the "quality of life" outcomes for Pakistan and Urdu speaking people.

DETAILED DESCRIPTION:
Data will be collected by PedQL Infants Scale Parent report A mix method approach will be applied Forward translation Backward translation Review of forward and backward translation The process of translation will be followed the guidelines in the translation manual. Translators will translate the PedsQL Inventory Infants Scale Parent Report independently from each other in Urdu language following the proper forward and backward translation procedure.

Data Analysis Quality of life pediatric population will assess through Urdu translated version of PedsQL Inventory Infants Scale Parent report. Data will be analyzed through SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Parents of both genders included
* Parents of infant age 1 to 12 months were included.

Exclusion Criteria:

* Parents suffering from psychological disorders
* Parents with severe behavior issue
* Parents who cannot understand Urdu

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample size was 43. Sample size was calculated by raosoft online software. Margin of error 5% Confidence level 95% Population size 20000 Response distribution 50% Sample Selection Criteria
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Quality of Life of Infants age 1 to 12 months | 6 months
  Urdu Translation and Cross Cultural Validation of PedsQL Inventory Infant Scale Parent Report 1 to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Saiqa Tabassum, MS, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah international university, Lahore, Punjab Province
  - Rising Sun Institute, Lahore, Punjab Province

REFERENCES:
- [Background] Varni JW, Limbers CA, Neighbors K, Schulz K, Lieu JE, Heffer RW, Tuzinkiewicz K, Mangione-Smith R, Zimmerman JJ, Alonso EM. The PedsQL Infant Scales: feasibility, internal consistency reliability, and validity in healthy and ill infants. Qual Life Res. 2011 Feb;20(1):45-55. doi: 10.1007/s11136-010-9730-5. Epub 2010 Aug 22. PMID 20730626